CLINICAL TRIAL: NCT04860908
Title: DOES COVID-19 INFECTION AND/OR VACCINATION OF PREGNANT WOMEN AFFECT THE PANCREATIC BETA CELLS OF THE FETUS BECOMING A TRIGGER FOR FUTURE DEVELOPMENT OF CHILDHOOD TYPE 1 DIABETES
Brief Title: COVID 19 ANTOBODIES IN PREGNANT WOMEN AND THEIR CONNECTION TO BETA CELL FUNCTION IN THE FETUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maaynei Hayesha Medical Center (Other)
Responsible Party: Principal Investigator, Mirra Manevich Mazor, OBSTETRICS & GYNECOLOGY RESIDENT, Maaynei Hayesha Medical Center
Other Study IDs: MaayneiHMC
Record Dates: First submitted 2021-04-26; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Generation of Anti COVID-19 Antibodies in a Fetus, Whose Mother Was Exposed to COVID or Was Vaccinated During Pregnancy
Keywords: covid-19 , antibodies, pregnancy, covid-19 vaccine, cord blood
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- covid exposed: women who were exposed to covid 19 during pregnancy
  Interventions: Other: no intervention, observation only
- covid vaccinated: women who were vaccinated to covid 19 during pregnancy
  Interventions: Other: no intervention, observation only

INTERVENTIONS:
Other: no intervention, observation only — no intervention, observation only

SUMMARY:
The aim of this study is to check for the presence of COVID 19 antibodies [Covid-19, GAD-65, IA-2, ICA] in the blood of laboring women who have been exposed to either the virus itself or to the vaccine during pregnancy . The same test will be done on cord blood. Then the types of antibodies will be compared, between maternal and neonatal blood. The blood will be taken along with routine blood tests without additional punctures of Mother or Baby.

DETAILED DESCRIPTION:
T1D is caused by an autoimmune reaction to proteins that cause the destruction of the pancreatic beta cells. The incidence of childhood Type 1 diabetes (T1D) is continuously increasing, caused by environmental factors, mainly viruses (1).

The most implicated viruses are coxsackie B4 (2) and rotaviruses (3,4). In the past mumps and rubella viruses gave been found to cause early childhood T1D and the introduction of mumps and rubella vaccination have stopped this process (5).

Recently we (6) and others (7-9) have shown that Rotavirus vaccination to infants attenuates the incidence of T1D in children aged 0-5 (in press). Covid-19 has not yet been investigated.

Aim of study To determine whether anti-Covid-19 antibodies generated by infection and/or vaccination of pregnant mothers, pass the placenta and affect the fetal beta-cells, by damaging or protecting these insulin producing cells.

Subjects 100 pregnant women with Covid-19 infection or vaccination who are followed and delivered at the Mayanei HaYeshua Medical Center will be enrolled in the study.

Method

Blood from the pregnant mothers will be taken at delivery (and before if possible) as well as from the cordblood. The following βcell specific antibodies will be tested in the laboratory of the Schneider Children's Hospital:

Covid-19, GAD-65, IA-2, ICA. (ml blood from the mother and 1ml cordblood) The bloods will have to be centrifuged within 20-30 minutes and the sera kept at -20ºC until delivery.

Background Whether the Covid-19 epidemic affects childhood T1D is controversial (10). Flannery et al (11) and Atyeo et al., reported that SARS-Cov-2 infected mothers transmit SARS-Cov-2 antibodies via the placenta to the fetus Fernandez reported protective Covid-19 antibodies in breast milk of infected mothers (13). Kamrath et al from Germany (14) and Rabbone et al from Italy (15) reported a high prevalence of DKA in children diagnosed with T1D during the recent pandemic.

As the Covid-19 virus with its various mutations is known to affect several organs and cells in the human body it is of great interest to know whether it affects also the pancreatic βcells of the fetus.

Hypothesis We assume that unvaccinated mothers transfer the virus antibodies to the fetus, and which may be the first damage to the βcells endangering future development of future type 1 childhood diabetes. Transfer of Covid protecting antibodies may beneficially affect the infant at risk.

Discussion and importance of the study To the best of our knowledge, no such study has been performed.

ELIGIBILITY:
Inclusion Criteria:

* exposure to the COVID 19 virus or vaccine during pregnancy

Exclusion Criteria:

- Age under 18 or over 48 IUFD

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — anyone with a uterus with a fetus in it may apply, gender identity not important
Study Population: pregnant women delivery a live infant who were exposed or vaccinated to COVID 19
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Presence of anti COVID 19 antibodies in maternal and cord blood | ONE YEAR
  Covid-19, GAD-65, IA-2, ICA

CONTACTS AND LOCATIONS:
Locations (1):
- Maayanei Hayeshua Medical Center, Bnei Brak, Central District, Israel

IPD SHARING:
Plan to Share IPD: Yes
IF YOU ASK NICELY WE'LL CONSIDER SHARING
Supporting Information: Study Protocol, ICF
Time Frame: ONE YEAR

REFERENCES:
- [Background] Op de Beeck A, Eizirik DL. Viral infections in type 1 diabetes mellitus--why the beta cells? Nat Rev Endocrinol. 2016 May;12(5):263-273. doi: 10.1038/nrendo.2016.30. Epub 2016 Mar 29. PMID 27020257